CLINICAL TRIAL: NCT01462305
Title: 30-Minute Light Exposure for the Treatment of Seasonal Affective Disorder
Acronym: SAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-1033-SADGO-MS
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Seasonal Affective Disorder
Keywords: SAD; Seasonal Affective Disorder; Winter Blues; Seasonal Depression
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- goLITE (Experimental): light therapy using 467nm LED source, within 30 minutes of waking in the morning every day for 6 weeks
  Interventions: Device: goLITE
- Control (Active Comparator): light therapy using 580nm LED source within 30 minutes of waking in the morning every day for 6 weeks
  Interventions: Device: Control

INTERVENTIONS:
Device: goLITE — goLITE at 30 minutes per day, within 30 minutes of waking in the morning
  Other Names: Light device; Blue Light
  Arms: goLITE
Device: Control — light therapy using 580nm LED source within 30 minutes of waking in the morning every day for 6 weeks
  Arms: Control

SUMMARY:
The primary objective of this study is to evaluate the effect of light therapy using a narrow 467nm light compared to a 580nm light in subjects with Seasonal Affective Disorder (SAD). It is hypothesized that the 467nm light will improve the symptoms of SAD better than the 580nm light.

DETAILED DESCRIPTION:
Participants will be randomly assigned to receive either a 467nm light or a 580nm light. Participants will use the light every day for six weeks for 30 minutes. Multiple assessments and questionnaires will be given weekly to assess the efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 21-64
2. Able and willing to provide written informed consent
3. History of recurrent major depressive episodes with winter-type seasonal pattern by Diagnostic and Statistical Manual of the American Psychiatric Associated, 4th Ed. (DSM-IV) criteria (American Psychiatric Association, 1990), based on diagnostic interview utilizing the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) (First et al., 2007)

   *Bipolar I excluded for this study
4. SIGH-ADS score of ≥20
5. Use of the light device as instructed by the study clinician for at least 6 out of 7 days for the first two weeks of therapy and at least 5 out of 7 days for the remaining four weeks of therapy.

Exclusion Criteria:

1. Participation in a study of investigational or marketed drugs or devices during the 30-day period prior to the start of the study or during the study
2. Subjects who are medically complicated, medically unstable and/or have other severe diseases, as determined by the investigator.
3. Abnormal TSH level, (outside range of 0.3 to 5.0 mlU/L), as determined by the TSH levels blood test
4. History of concurrent psychiatric illness that would preclude compliance with the protocol and/or ability to complete the study safely
5. History or current diagnosis of Bipolar I Disorder
6. Variable psychiatric symptoms such as rapid cycling or severe premenstrual syndrome that could interfere with accurate assessment of the treatment effect
7. History of a medical condition that affects mood or produces hallmark symptoms of a mood disorder (i.e. hypothyroidism)
8. History of current or recent (within previous 12 months) alcohol, narcotic or other drug abuse by DSM-IV criteria
9. Positive urine drug screen at the Physical Screening
10. Active suicidal or homicidal ideation or plan, as determined by the investigator
11. Global Assessment of Functioning (GAF) <51 (see Appendix B)
12. Use of light therapy treatment within the previous 6 months or any history of goLITE use
13. Pregnant or lactating (will confirm absence of pregnancy with a urine or serum pregnancy test in females of childbearing potential during the Physical Screening. Additional pregnancy tests may be performed as per individual site requirements). Females of child-bearing potential must agree to use some form of birth control throughout the course
14. Current use or use within 2 months of antidepressants or mood stabilizing medications, even if taken for a non-psychiatric indication
15. Currently working night shift or rotating shift or other habitual alteration of the sleep/wake cycle
16. Planned travel outside of the state in which the trial is being conducted
17. Current use or use within the previous 1 month of photosensitizing medications (amiodarone, benoxaprofen, chlorpromazine, demeclocycline, fleroxacin, nalidixic acid, ofloxacin, piroxicam, porfimer, psoralens, quinidine, temoporfin) or remedies (St. John's wort, melatonin)
18. History of eye trauma or disease, retinopathy, and/or cataract of a level that would significantly affect transmission or processing of light through either eye
19. Ishihara score of <10 on the Ishihara Test for Color Deficiency
20. Use of medications, such as tetracycline or oral isoretinoin (Accutane), that would affect the safety of light exposure treatment or that causes complaints of eyestrain or abnormal tearing with computer use of up to 30 minutes at a time

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2012-04-02 (Actual); Study Completion 2012-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Anderson, PhD, Principal Investigator — Brigham and Women's Hospital; Robert Auger, MD, Principal Investigator — Mayo Clinic; Scott Crow, MD, Principal Investigator — University of Minnesota; Carol Glod, PhD, Principal Investigator — Mclean Hospital; Alfredo Rivera, MD, Principal Investigator — Community Research Management Associates
Locations (4):
- United States (4):
  - McLean Hospital, Belmont, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Community Research Management Associates, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects in this multicenter trial were recruited and treated at one of five participating sites between January and March 2012. Fifty-six subjects were recruited from 5 health care centers. Twenty-one failed to meet all the inclusion/exclusion criteria, including depression severity and were not randomized into the study.
Period: Overall Study
Arm/Group | goLITE | Control
Started | 18 | 17
Completed | 16 | 13
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | goLITE | Control | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11.1) | 38.9 (11.4) | 44.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: SIGH-ADS Score
Description: A Structured Interview Guide for the Hamilton Depression Scale with Atypical Depression Supplement was utilized at baseline and after 6 weeks of treatment.
  The SIGH-ADS is designed for general use in depression research and clinical evaluation, regardless of seasonality.The SIGH-ADS rates the severity of depressive symptoms in terms of Hamilton's 17-item depression score and an 8-item atypical score. Combined this provides 25 items to provide the SIGH-ADS score. SIGH-ADS scores range from 0-79; higher values represent increased depression severity and worse outcome, the lower the score the less depressed the patient is. All participants that entered the study had to have a score of 20 or greater.
Time Frame: 6 weeks
Population: Of the 35 participants that were randomized 29 completed the study the SIGH-ADS at week 6.
  3 subjects withdrew due to treatment-related adverse events 3 withdrew for non-study-related reasons.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | goLITE | Control
Number analyzed (Participants) | 18 | 17
units on a scale
  Baseline | 29.4 (5.3) | 25.8 (5.1)
  Week 6: number analyzed (Participants) | 16 | 13
  Week 6 | 5.6 (6.1) | 4.5 (5.3)
Statistical Analysis 1: Comparison: goLITE vs Control; To test the hypothesis that depressed SAD patients would demonstrate greater antidepressant therapeutic benefit from the ~465nm (shorter wavelength) source compared with the ~595nm (longer wavelength) source, we conducted a repeated-measures ANOVA using PROC MIXED in SAS 9.3 with treatment (~465nm vs. ~595nm) as a between-subject factor and time (treatment visit 1, treatment visit 2, treatment visit 3, phone assessment 1, phone assessment 2, and treatment visit 4) as a within-subject factor; Test type: Superiority or Other; p = 0.74, ANOVA — interaction effect and week of treatment condition
Statistical Analysis 2: Comparison: goLITE vs Control; Test type: Superiority or Other; p = 0.9, ANOVA — A repeated-measures ANOVA on the 29 subjects revealed no significant effect or interaction effect
Statistical Analysis 3: Comparison: goLITE vs Control; Test type: Superiority or Other; p < 0.0001, ANOVA — A repeated-measures ANOVA on the 29 subjects revealed significant effect of treatment week

2. Secondary Outcome: SIGH-ADS Score (Week 1 Thru 5)
Description: A Structured Interview Guide for the Hamilton Depression Scale with Atypical Depression Supplement was utilized weekly at in person visits or over the phone.
  The SIGH-ADS is designed for general use in depression research and clinical evaluation, regardless of seasonality.The SIGH-ADS rates the severity of depressive symptoms in terms of Hamilton's 17-item depression score and an 8-item atypical score. Combined this provides 25 items to provide the SIGH-ADS score. SIGH-ADS scores range from 0-79; higher values represent increased depression severity and worse outcome and the lower the score the less depressed the patient is. All participants that entered the study had to have a score of 20 or greater.
Time Frame: weekly, from Week 1 through week 5
Population: Of the 35 participants that were randomized 29 completed the study the SIGH-ADS at week 6.
  3 subjects withdrew due to treatment-related adverse events 3 withdrew for non-study-related reasons. Not all participants were able to complete the study related site visits or phone calls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | goLITE | Control
Number analyzed (Participants) | 17 | 14
units on a scale
  Week 1 | 17.3 (9.6) | 16.9 (7.5)
  Week 2: number analyzed (Participants) | 16 | 14
  Week 2 | 14.4 (8.7) | 13.7 (8.3)
  Week 3: number analyzed (Participants) | 16 | 14
  Week 3 | 12.1 (7.0) | 9.3 (8.6)
  Week 4 (phone call): number analyzed (Participants) | 15 | 13
  Week 4 (phone call) | 10.2 (7.4) | 6.7 (6.5)
  Week 5 (phone call): number analyzed (Participants) | 14 | 13
  Week 5 (phone call) | 7.6 (5.9) | 5.5 (5.6)

3. Secondary Outcome: Q-LES-Q-SF
Description: The Q-LES-Q-SF (Quality of life enjoyment and satisfaction questionnaire short form) is a 16 question questionnaire that is enables investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning.
  Responses to questions range from 1 to 5, 1 being very poor and 5 being very good. Scores range from 16 to 80, the higher score the higher the participants enjoyment and satisfaction.
Time Frame: 6 weeks
Population: Of the 35 participants that were randomized 28 completed the Q-LES-Q-SF at week 6.
  3 subjects withdrew due to treatment-related adverse events 3 withdrew for non-study-related reasons.
  Not all participants were able to complete the study related site visits or phone calls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | goLITE | Control
Number analyzed (Participants) | 15 | 16
units on a scale
  Baseline | 42.5 (7.1) | 43.6 (6.4)
  Week 3: number analyzed (Participants) | 15 | 12
  Week 3 | 51.1 (6.3) | 52.2 (7.3)
  Week 6: number analyzed (Participants) | 15 | 13
  Week 6 | 55.3 (9.9) | 57.0 (7.8)
Statistical Analysis 1: Comparison: goLITE vs Control; Test type: Superiority or Other; p = 0.20, ANOVA

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | goLITE | Control
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 12/18 | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | goLITE (N=18) | Control (N=17)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 7 (10)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 (2) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Eye Sensitivity (Eye disorders) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 3 (4)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
nasal sinus irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
cold (Immune system disorders) | 4 (4) | 3 (3)
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
backache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sinus infection (Infections and infestations) | 1 (1) | 0 (0)
hot spot on eye (Eye disorders) | 1 (1) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
eye strain (Eye disorders) | 1 (1) | 1 (1)
facial warming (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GI upset (Gastrointestinal disorders) | 1 (1) | 0 (0)
itchy/watery eyes (Eye disorders) | 1 (1) | 0 (0)
perimenstrual symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1) — perimenstrual headache and cramps
white flashing lights (Eye disorders) | 0 (0) | 1 (1)
bloody nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No